CLINICAL TRIAL: NCT02736123
Title: Neoadjuvant Combination Biotherapy With Ipilimumab and Nivolumab or Nivolumab Alone in Patients With Locally/Regionally Advanced/Recurrent Melanoma: A Randomized Efficacy, Safety and Biomarker Study
Brief Title: Neoadjuvant Combination Biotherapy With Ipilimumab and Nivolumab or Nivolumab Alone
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: PI is closing the trial as he will be leaving the University of Pittsburgh Medical Center
Sponsor: University of Pittsburgh (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Ahmad Tarhini, Principal Investigator, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15-113
Record Dates: First submitted 2016-03-28; First posted 2016-04-13 (Estimated); Last update posted 2017-09-20 (Actual); Status verified 2017-09

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A consists of 3 phases or steps (Experimental): Induction Phase Nivolumab 3 mg/kg IV infusion every 2 weeks for 3 doses
  Definitive Surgery Complete lymph node dissection/ lymphatic, cutaneous, subcutaneous disease resection (week 6-8+)
  Maintenance Phase (after recovery from surgery) Nivolumab 3 mg/kg IV infusion every 3 weeks
  Interventions: Drug: Nivolumab - Arm A
- Arm B consists of 3 phases or steps (Experimental): Nivolumab 1 mg/kg IV infusion every 3 weeks for 2 doses given concurrently with Ipilimumab 3 mg/kg IV infusion every 3 weeks for 2 doses
  Definitive Surgery Complete lymph node dissection/ lymphatic, cutaneous, subcutaneous disease resection (week 6-8+)
  Maintenance Phase (after recovery from surgery) Nivolumab 1 mg/kg IV infusion every 3 weeks for 2 doses given concurrently with Ipilimumab 3 mg/kg IV infusion every 3 weeks for 2 doses; then, Nivolumab 3 mg/kg IV infusion every 3 weeks
  Interventions: Drug: Nivolumab + Ipilimumab - Arm B

INTERVENTIONS:
Drug: Nivolumab - Arm A — Nivolumab will be given during the induction phase of the study for 6 weeks. This is followed by surgery. Then maintenance therapy (after recovery from surgery).
  Arms: Arm A consists of 3 phases or steps
Drug: Nivolumab + Ipilimumab - Arm B — Nivolumab + ipilimumab during the induction phase of the study for 6 weeks. This is followed by surgery (week 6-8+). Then maintenance therapy will be initiated for up to one year from study drug initial administration ((after recovery from surgery).
  Arms: Arm B consists of 3 phases or steps

SUMMARY:
This study plans to test the pathologic complete response (pCR) rate of the combination biotherapy regimen consisting of nivolumab plus ipilimumab versus nivolumab alone in patients with advanced but operable melanoma. Evaluation of the presence of tumor-infiltrating CD8+ T cells as well as that of PDL1 expression and IDO expression will be associated with clinical response (pathologic and/or radiologic). The study will test the radiologic/clinical preoperative response rate, recurrence free survival (RFS) and overall survival (OS). It will evaluate the safety of neoadjuvant nivolumab and neoadjuvant nivolumab-ipilimumab. Up to 66 patients will be randomized in 1:1 ratio.

DETAILED DESCRIPTION:
The study has 2 study arms:

* Nivolumab alone (Arm A)

  * Induction phase: nivolumab 3 mg/kg IV infusion every 2 weeks x3 doses. Followed by Definitive Surgery.
  * Maintenance phase: nivolumab 3 mg/kg IV infusion every 3 weeks for up to one year from study treatment initiation.
* Ipilimumab + nivolumab (Arm B)

  * Induction phase: Ipilimumab 3 mg/kg IV + Nivolumab 1 mg/kg IV every 3 weeks x2. Followed by Definitive Surgery.
  * Maintenance phase: nivolumab 3 mg/kg IV infusion every 2 weeks for up to one year from study treatment initiation.

Definitive Surgery consists of complete lymph node dissection/ lymphatic, cutaneous, subcutaneous or other distant disease resection (week 6-8+).

ELIGIBILITY:
Inclusion Criteria:

* Men and women at least 18 years of age
* Willing and able to give written informed consent
* Performance status Eastern Cooperative Oncology Group (ECOG) zero or 1
* Histologic diagnosis of melanoma belonging to the following AJCC Tumor Node and Metastasis (TNM) stages: Tx or T1-4 and N1b or N2 or N2c or N3 and/or M0 or M1 (if considered surgically operable)
* Patients are eligible for this trial either at presentation for primary melanoma with concurrent regional nodal and/or in-transit metastasis and/or distant metastasis, or at the time of clinically detected nodal and/or in-transit recurrence and/or distant metastasis and may belong to any of the following groups: Primary melanoma with clinically apparent (overt) regional lymph node metastases.
* Clinically detected recurrence of melanoma at the proximal regional lymph node(s) basin.
* Clinically detected primary melanoma involving multiple regional nodal groups.
* Clinically detected site of nodal metastatic melanoma arising from an unknown primary.
* Patients with intransit or satellite metastases with or without lymph node involvement are allowed if they are considered surgically resectable at baseline.
* Patients with distant metastases with or without intransit or lymph node involvement are allowed if they are considered potentially surgically resectable at baseline. NOTE: All patients must be determined to be surgically resectable at baseline to be eligible for this neoadjuvant study.
* Have measurable disease based on RECIST 1.1.
* Have provided tumor tissue from a newly obtained core, punch, incisional or excisional tumor biopsy. Patients must undergo biopsy (core, punch) or open incisional/excisional biopsy (if done as part of a clinically indicated baseline diagnostic procedure) within 4 weeks of registration on the study.
* Patients must have been evaluated by standard-of-care full body imaging studies (CT, PET/CT or MRI) as part of the initial clinical work-up at baseline (no more than 4 weeks prior to study enrollment) and after completion of induction nivolumab-ipilimumab or nivolumab alone (at 6-8 weeks after the first dose of induction and prior to the definitive surgery procedure).
* Required values for initial laboratory tests:

  * White blood cell (WBC) 3000/uL
  * Absolute neutrophil count (ANC) 1500/uL
  * Platelets 100 x 103/uL
  * Hemoglobin 10 g/dL
  * Aspartate transaminase/alanine transaminase (AST/ALT) 2.5 x unique learner number (ULN)
  * Bilirubin 1.5 ULN, (except patients with Gilbert's Syndrome, who must have a total bilirubin less than 3.0 mg/dL)
  * Serum creatinine ≤ 1.5 x ULN or creatinine clearance (CrCl) ≥ 40 mL/min (if using the Cockcroft-Gault formula below):

Female CrCl = (140 - age in years) x weight in kg x 0.85 72 x serum creatinine in mg/dL Male CrCl = (140 - age in years) x weight in kg x 1.00 72 x serum creatinine in mg/dL

• No active or chronic infection with HIV, Hepatitis B, or Hepatitis C

Exclusion Criteria:

* Subject will be excluded from participating in the trial if they meet any of the following criteria:
* Patients are excluded if they have a history of central nervous system (CNS)metastases.
* Patients who have had a history of acute diverticulitis, intra-abdominal abscess, GI obstruction and abdominal carcinomatosis which are known risk factors for bowel perforation.
* Any other malignancy from which the patient has been disease-free for less than 3 years, with the exception of adequately treated and cured basal or squamous cell skin cancer, superficial bladder cancer or carcinoma in situ of the cervix.
* Patients will be excluded if they have an active, known or suspected autoimmune disease. Autoimmune disease: Patients with a history of inflammatory bowel disease are excluded from this study, as are patients with a history of symptomatic autoimmune disease (e.g., rheumatoid arthritis, systemic progressive sclerosis (scleroderma), systemic lupus erythematosus, autoimmune vasculitis e.g., Wegener's Granulomatosis); motor neuropathy considered of autoimmune origin (e.g. Guillain-Barre Syndrome).
* Subjects are permitted to enroll if they have vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger.
* Has evidence of interstitial lung disease or active, non-infectious pneumonitis.
* Patients should be excluded if they have a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.
* As there is potential for hepatic toxicity with nivolumab or nivolumab/ipilimumab combinations, drugs with a predisposition to hepatoxicity should be used with caution in patients treated with nivolumab-containing regimen.
* Has an active infection requiring systemic therapy.
* Has received a live vaccine within 30 days prior to the first dose of trial treatment.
* Any underlying medical or psychiatric condition, which in the opinion of the Investigator/Sub-Investigator will make the administration of ipilimumab or nivolumab hazardous or obscure the interpretation of adverse events (AEs), such as a condition associated with frequent diarrhea.
* Patients with underlying heart conditions who are deemed ineligible for surgery by cardiology consult.
* A history of prior treatment with ipilimumab, nivolumab or other cytotoxic T-lymphocyte-associated protein (CTLA-4), progressive disease (PD1) or PD-L1 inhibitor.
* Prior treatment with interferon alfa is allowed.
* A history of prior radiotherapy, chemotherapy, including infusion or perfusion therapy for current disease or any immunotherapy including tumor vaccines, interferon-alfa, interleukins, levamisole or other biologic response modifiers within the past 4 weeks.
* Concomitant therapy with any of the following: IL 2 or other non-study immunotherapy regimens; cytotoxic chemotherapy; immunosuppressive agents; other investigation therapies; or chronic use of systemic corticosteroids; unless discontinued ≥ 4 weeks. A history of occasional use of steroid inhalers is allowed.
* Women of childbearing potential (WOCBP), defined above in Section 3.3, who are unwilling or unable to use an acceptable method of contraception to avoid pregnancy for their entire study period and for at least 23 weeks after cessation of study drug, or have a positive pregnancy test at baseline, or are pregnant or breastfeeding.
* Melanoma of Uveal Origin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-10; Primary Completion 2017-02-09 (Actual); Study Completion 2017-02-09 (Actual)

PRIMARY OUTCOMES:
Assess the pathologic complete response rate (absence of viable tumor on histologic assessment) | 5 years

SECONDARY OUTCOMES:
Evaluate preoperative clinical/radiologic response rate | 5 years
Assess progression free survival | 5 years
Assess overall survival | 5 years
Assess biomarkers CD8 T cell, PD-L1 and IDO expression by immunohistochemistry | 5 years
Assess safety and adverse events | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad Tarhini, MD, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Cancer Center Hillman Cancer Center, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] Gorry C, McCullagh L, O'Donnell H, Barrett S, Schmitz S, Barry M, Curtin K, Beausang E, Barry R, Coyne I. Neoadjuvant treatment for stage III and IV cutaneous melanoma. Cochrane Database Syst Rev. 2023 Jan 17;1(1):CD012974. doi: 10.1002/14651858.CD012974.pub2. PMID 36648215